CLINICAL TRIAL: NCT04968691
Title: Investigation of Results of Structured Exercise Application Based on Telerehabilitation in Individuals With Unilateral Transtibial Amputation
Brief Title: Telerehabilitation in Individuals With Unilateral Transtibial Amputation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mehmet Kurtaran (Other)
Responsible Party: Sponsor-Investigator, Mehmet Kurtaran, Principal Investigator, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-15
Record Dates: First submitted 2021-07-07; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Amputation; Telerehabilitation; Exercise; Prosthesis User
Keywords: Transtibial Amputation; Below Knee Amputation; Transtibial Prosthesis Users; Below Knee Prosthesis Users; Telerehabilitation; Amputees Rehabilitation; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): The group to which a structured exercise program supported by telerehabilitation will be treated.
  Interventions: Other: Telerehabilitation based exercise treatment
- Control group (Active Comparator): The group to which the home exercise program will be treated.
  Interventions: Other: Home based exercise treatment

INTERVENTIONS:
Other: Telerehabilitation based exercise treatment — The telerehabilitation group will be shown how to do the exercises online by the researcher before each session, 3 sessions a week for 6 weeks, with mobile telecommunication applications, and it will be ensured that the patients do the exercises correctly and are followed up. In addition, at the beginning of each week, videos with the exercise content of that week will also be sent.
  Arms: Telerehabilitation group
Other: Home based exercise treatment — n the study, exercise cards were given to the control group and the exercise treatment they were asked to do at home 3 sessions a week for 6 weeks
  Arms: Control group

SUMMARY:
It is aimed to investigate the effects of telerehabilitation-based structured exercise on muscle strength, balance, performance, body image, prosthesis adaptation, activity limitation, prosthesis use satisfaction, and quality of life in individuals with unilateral below-knee amputation. Study hypothesis: In individuals with transtibial amputation, telerehabilitation-based structured exercise has an effect on muscle strength, balance, performance, body image, prosthesis adaptation, activity limitation, prosthesis use satisfaction, and quality of life. Forty individuals with a unilateral transtibial amputation will be included in the study. Participants will be divided into two groups as telerehabilitation and control groups with equal sample sizes by the randomization method. All participants will undergo a 6-week exercise program. A structured exercise program supported by telerehabilitation will be applied to the telerehabilitation group 3 days a week, and a home exercise program will be applied on the remaining days of the week. An only a home exercise program will be applied to the control group. Participants will be evaluated at the beginning and end of the study.

DETAILED DESCRIPTION:
Amputation is a major trauma that significantly disrupts the biomechanics of the musculoskeletal system, results in serious physical and psychological loss, and completely affects the quality of life, social and professional life of the individual. Due to the increase in the elderly population and the incidence of diabetes and vascular diseases in the world, the number of individuals with amputation is increasing day by day. Approximately 150,000 lower extremity amputations are performed each year in the United States alone. The number of amputated individuals worldwide is expected to double by 2050. The most common amputation level in the world and in our country is transtibial amputations and approximately 39% of all amputations are performed at this level. In addition, the most common prosthesis use among individuals with lower extremity amputations is seen in those with the transtibial amputation level. Individuals who have undergone transtibial amputation have lost the foot-ankle complex and all related muscular functions. After transtibial amputation surgery, loss of proprioceptive information occurs in ankle control and in foot-ankle and all lower extremity muscles due to loss of exteroceptors around the foot. This leads to loss of balance during standing, stepping, and walking.

Physiotherapy and rehabilitation practices are needed in order for individuals with amputations to use their prostheses effectively and have a successful prosthesis adaptation. After the transtibial amputation, early period physiotherapy applications are followed by the use of prosthesis, and prosthetic period rehabilitation applications are continued. Prosthetic rehabilitation in individuals with transtibial amputation; aims to provide balance by taking into account the losses after amputation, to gain close to normal walking with minimum energy consumption, to ensure maximum independence in a safe manner by taking into account the pre-amputation lifestyles, expectations, and medical limitations of individuals. Physiotherapy and rehabilitation practices in individuals with transtibial amputation consist of a long-term process that starts before amputation and includes the early period after amputation, the prosthetic period, and returns to social life. Factors such as the long-term physiotherapy needs of individuals with transtibial amputation, the presence of gait and balance problems, geographical conditions, financial inadequacies, and epidemic diseases may cause problems for these individuals to reach the physiotherapy and rehabilitation applications offered in health institutions. In order to facilitate participation in physiotherapy and rehabilitation practices and to reduce resource use, telerehabilitation practices are recommended for individuals with amputation, as with other diseases that require rehabilitation. It is thought that telerehabilitation can be a useful and practical method for individuals with transtibial amputation where it is difficult and tiring to go to the clinic.

In the literature, it has been observed that there are very few studies examining the effects of physiotherapy and rehabilitation on parameters such as muscle strength, balance, gait, performance, body image, prosthesis fit, prosthesis use satisfaction, and quality of life in the rehabilitation of individuals with transtibial amputation. In addition, there are very few studies in the literature that include telerehabilitation applications related to transtibial amputations, and there is no study that questions the effects of structured exercise programs. This study was planned in order to determine the effects of telerehabilitation applications on muscle strength, kinesiophobia, balance, activity limitation, body image, prosthesis compliance and satisfaction with use, and quality of life in individuals with transtibial amputation. It is aimed to guide physiotherapists whether they prefer telerehabilitation applications as an evidence-based practice among rehabilitation methods in this field.

It is aimed to investigate the effects of telerehabilitation-based structured exercise on muscle strength, balance, performance, body image, prosthesis adaptation, activity limitation, prosthesis use satisfaction, and quality of life in individuals with unilateral transtibial amputation.

In order to determine the number of samples in the study; the alpha significance level of the hypothesis was 0.05; the effect size was determined as 0.5 and power as 0.85. As a result of the analysis; The research will be carried out with a total of 40 people, 20 people in each group.

Forty individuals with a unilateral transtibial amputation will be included in the study. Participants will be divided into two groups as telerehabilitation and control groups with equal sample sizes by the randomization method. All participants will undergo a 6-week exercise program. A structured exercise program supported by telerehabilitation will be applied to the telerehabilitation group 3 days a week, and a home exercise program will be applied on the remaining days of the week. An only a home exercise program will be applied to the control group. Participants will be evaluated at the beginning and end of the study.

Method of the Study:

* A mobile telecommunication group will be formed, including the participants and the physiotherapist. Communication with the participants will be provided here. In addition, one-on-one or collective teleconferences will be held with the participants when necessary.
* Before each session, the telerehabilitation group will be shown how to do the exercises online by the researcher, and it will be ensured that the patients do the exercises correctly and are followed up. In addition, at the beginning of each week, videos with the exercise content of that week will also be sent.
* The control group will be given exercise cards showing the home exercise program at the beginning of the treatment.
* Tracking of the exercises will be done with the exercise diary Statistical analysis: In the analysis of the data, statistical analysis including a descriptive, comparator, and correlation will be made. Mean, standard deviation and percentage distributions will be calculated for descriptive data. In the analysis of the repeated measurement results of the scales, ANOVA will be applied for the data conforming to the normal distribution. The student's t-test will be used for parametric data and Mann Whitney-U test for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Having a unilateral transtibial amputation
* Using active vacuum system prosthesis and carbon foot for at least one year
* Being at the level of mobility level K2-K3
* Not having any problems in the healthy leg
* A score of 21 or higher on the Montreal cognitive assessment scale (MOCA)

Exclusion Criteria:

* Patients who received physical therapy in the last 6 months
* Having a neurological, orthopedic, and systemic condition that will prevent them from exercising
* Having any orthopedic and neurological problems in the upper extremity
* Having severe hearing, vision, and speech impairment

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The Timed Up and Go test | up to 20 weeks
  The Timed Up and Go test is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require.
30 Second Sit to Stand Test | up to 20 weeks
  lso known as a 30-second chair stand test, this test is a way to assess an individual's leg strength and endurance by having them stand up from a sitting position repeatedly over the course of 30 seconds.

SECONDARY OUTCOMES:
Trinity Amputation and Prosthesis Experiences Scales (TAPES) | up to 20 weeks
  TAPES consists of 9 subscales. There are 3 psychosocial subscales: general adjustment , social adjustment, and adjustment to limitation. Scores range from 5 to 25, with higher scores indicating greater levels of adjustment. The TAPES also contain 3 activity restriction subscales: functional activity restriction , social activity restriction , and athletic activity restriction . Scores range from 3 to 12, with higher scores indicating greater activity restriction. There are 3 additional subscales that assess satisfaction with the prosthesis, measured along a 5-point scale (very dissatisfied, dissatisfied, neither dissatisfied nor satisfied, satisfied, very satisfied). Higher scores in each of the satisfaction subscales indicate greater satisfaction with the prosthesis.
Activities-specific Balance Confidence Scale (ABC Scale) | up to 20 weeks
  The ABC scale contains 16 tasks related to indoor and outdoor daily living activities, to measure balance confidence in elderly people who have various levels of functioning. Scores range from 0% (no confidence) to 100% (complete confidence) for each question item. Higher scores indicate greater confidence.

OTHER OUTCOMES:
The Amputee Body Image Scale (ABIS) | up to 20 weeks
  ABIS is comprised of 20 items. The response to each item ranges from 1 (none of the time) to 5 (all of the time). This scale produces scores that range from 20-100, with high scores indicating high body image disturbance. Three questions (question 3, 12 and 16) are reverse-scored.
The Nottingham Health Profile | up to 20 weeks
  The Nottingham Health Profile (NHP) is a general patient-reported outcome measure which seeks to measure subjective health status. It is a questionnaire designed to measure a patient's view of their own health status, in a number of areas. The NHP consists of two parts. The first part focuses on health and comprises 38 items which deal with pain, energy, sleep, mobility, emotional reaction and social isolation. The second part focuses on life areas affected and consists of 7 items which deal with problems regarding occupation, housework, social life, family life, sexual function, hobbies and holidays. Scoring is straightforward, with 0 assigned to a 'no' response and 1 to a 'yes' response. Scores for each of the sections range between 0 ('worst health') and 100 ('best health').

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kurtaran, MSc, Principal Investigator — Istanbul Universtiy- Cerrahpasa; Derya Çelik, PhD, Study Director — Istanbul Universtiy- Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa Faculty of Health Science, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All IPD that underlie results will not be shared

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Highsmith MJ, Kahle JT, Miro RM, Orendurff MS, Lewandowski AL, Orriola JJ, Sutton B, Ertl JP. Prosthetic interventions for people with transtibial amputation: Systematic review and meta-analysis of high-quality prospective literature and systematic reviews. J Rehabil Res Dev. 2016;53(2):157-84. doi: 10.1682/JRRD.2015.03.0046. PMID 27149143
- [Background] Davie-Smith F, Paul L, Nicholls N, Stuart WP, Kennon B. The impact of gender, level of amputation and diabetes on prosthetic fit rates following major lower extremity amputation. Prosthet Orthot Int. 2017 Feb;41(1):19-25. doi: 10.1177/0309364616628341. Epub 2016 Jul 9. PMID 26850990
- [Background] Dillingham TR, Pezzin LE, Shore AD. Reamputation, mortality, and health care costs among persons with dysvascular lower-limb amputations. Arch Phys Med Rehabil. 2005 Mar;86(3):480-6. doi: 10.1016/j.apmr.2004.06.072. PMID 15759232
- [Background] Hsu MJ, Nielsen DH, Lin-Chan SJ, Shurr D. The effects of prosthetic foot design on physiologic measurements, self-selected walking velocity, and physical activity in people with transtibial amputation. Arch Phys Med Rehabil. 2006 Jan;87(1):123-9. doi: 10.1016/j.apmr.2005.07.310. PMID 16401450
- [Background] Hofstad CJ, van der Linde H, Nienhuis B, Weerdesteyn V, Duysens J, Geurts AC. High failure rates when avoiding obstacles during treadmill walking in patients with a transtibial amputation. Arch Phys Med Rehabil. 2006 Aug;87(8):1115-22. doi: 10.1016/j.apmr.2006.04.009. PMID 16876558
- [Background] Broomhead P, Clark K, Dawes D, Hale C, Lambert A, Quinlivan D, et al. Evidence-based clinical guidelines for the physiotherapy management of adults with lower limb prostheses. Chartered Society of Physiotherapy. 2012, 2nd. London.
- [Background] Rintala DH, Krouskop TA, Wright JV, Garber SL, Frnka J, Henson HK, Itani KM, Gaddis W, Matamoros R, Monga TN. Telerehabilitation for veterans with a lower-limb amputation or ulcer: Technical acceptability of data. J Rehabil Res Dev. 2004 May;41(3B):481-90. doi: 10.1682/jrrd.2004.03.0481. PMID 15543466
- [Background] Nelson VS, Flood KM, Bryant PR, Huang ME, Pasquina PF, Roberts TL. Limb deficiency and prosthetic management. 1. Decision making in prosthetic prescription and management. Arch Phys Med Rehabil. 2006 Mar;87(3 Suppl 1):S3-9. doi: 10.1016/j.apmr.2005.11.022. PMID 16500187
- [Background] Jones CJ, Rikli RE. Measuring functional fitness of older adults. J Active Aging. 2002; 24-30.
- [Background] Ayhan Ç, Büyükturan Ö, Kırdı N, Yakut Y, Güler Ç. The Turkish vercion of the Activites Specific Balance Confidence (ABC) Scale: Its cultural adaptation, validation and reliability in older adults. Turkish Journal of Geriatrics, 2014;17(2),157-163.
- [Background] Topuz S, Ulger O, Yakut Y, Gul Sener F. Reliability and construct validity of the Turkish version of the Trinity Amputation and Prosthetic Experience Scales (TAPES) in lower limb amputees. Prosthet Orthot Int. 2011 Jun;35(2):201-6. doi: 10.1177/0309364611407678. PMID 21697202
- [Background] Bumin G, Bayramlar K, Yakut Y, Sener GY. Cross cultural adaptation and reliability of the Turkish version of Amputee Body Image Scale (ABIS). J Back Musculoskelet Rehabil. 2009;22(1):11-6. doi: 10.3233/BMR-2009-0208. PMID 20023358
- [Background] Demet K, Guillemin F, Martinet N, Andre JM. Nottingham Health Profile: reliability in a sample of 542 subjects with major amputation of one or several limbs. Prosthet Orthot Int. 2002 Aug;26(2):120-3. doi: 10.1080/03093640208726634. PMID 12227446
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273